CLINICAL TRIAL: NCT01767545
Title: Twelve Months Experience With a Dexamethasone-implant for the Treatment of Macular Edema Associated With Retinal Vein Occlusion
Brief Title: Dexamethasone-implant for the Treatment of RVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Wolfgang Mayer, MD, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Mayer-DEX-001
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Macular Edema Caused by Retinal Vein Occlusion
MeSH Terms: interventions — Dexamethasone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone-implant (Group 1) (Active Comparator): Group 1 included 38 patients (22 with CRVO and 16 with BRVO) and was treated with a dexamethasone-implant injection from the beginning.
  Interventions: Drug: Dexamethasone implant
- Bevacizumab/Dexamethasone-implant (Group 2) (Active Comparator): Group 2 included 26 patients (14 CRVO, 12 BRVO) and was treated with three consecutive injections of bevacizumab at a monthly interval, followed by a dexamethasone-implant injection four weeks after the last bevacizumab injection.
  Interventions: Drug: Dexamethasone implant; Drug: Bevacizumab

INTERVENTIONS:
Drug: Dexamethasone implant
Drug: Bevacizumab
  Arms: Bevacizumab/Dexamethasone-implant (Group 2)

SUMMARY:
To evaluate the efficacy and safety of a dexamethasone-implant alone or in combination with bevacizumab. 64 eyes are prospectively investigated. Group 1 (22 CRVO and 16 BRVO) is treated with dexamethasone-implant alone, Group 2 (14 CRVO 12 BRVO) with three consecutive bevacizumab injections followed by a dexamethasone-implant. Recurrences are treated with dexamethasone-implant only. Patients are seen preoperatively and thereafter in monthly intervals. The primary endpoint was BCVA at twelve months.

ELIGIBILITY:
Inclusion Criteria: maximum duration of symptoms of four months and no known history of glaucoma or corticosteroid response in the past -

Exclusion Criteria: Glaucoma, Diabetic Retinopathy, prior IVOM, Uveitis

-

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary clinical endpoint was BCVA twelve months after the first intravitreal treatment. | 12 months

SECONDARY OUTCOMES:
Central retinal thickness | 12 months
Lens opacity | 12 months
Saftey of procedure | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Ophthalmology, LMU Munich, Munich, Germany